CLINICAL TRIAL: NCT00393120
Title: A Randomized, Double-blind, Placebo-controlled Study Exploring the Safety, Tolerability, PK & Virological Effect of Once Daily Oral Dosing of INCB009471 as Monotherapy for 14 Days in ARV-naïve/Limited ARV-experienced, HIV-1 Infected Pts.
Brief Title: Safety/Effectiveness of Oral Chemokine Coreceptor 5 (CCR5) Antagonist INCB009471 in R5-tropic HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Rich Levy, MD, Incyte Corporation
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 9471-201; INCB 9471-201 (Other: Incyte Corporation); IND No.69,030
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: HIV Infections
Keywords: HIV-infection; viral load; CCR5; viral tropism; HIV-1 infection; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A - INCB009471 100mg IR (Experimental): INCB009471, 100 mg IR orally once daily
  Interventions: Drug: INCB009471
- Treatment B - INCB009471 300mg SR (Experimental): INCB009471, 300 mg SR orally once daily
  Interventions: Drug: INCB009471
- Treatment C - Placebo (Placebo Comparator): Placebo matching INCB009471
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: INCB009471 — 100mg SR (sustained release) orally once daily
  Arms: Treatment A - INCB009471 100mg IR
Drug: INCB009471 — 300mg SR (sustained release) orally once daily
  Arms: Treatment B - INCB009471 300mg SR
Drug: Placebo comparator — Orally once daily
  Arms: Treatment C - Placebo

SUMMARY:
This study will evaluate the safety, pharmacokinetics and efficacy of the CCR5 antagonist INCB009471 in HIV-1 infected patients who are antiretroviral therapy naïve, or who are not currently on a HAART regimen and have not received any antiretroviral agents for 3 months prior to the Screening visit. Subjects will receive study medication (INCB009471) admnistered orally or placebo once daily with food for 14 days. Clinical safety laboratories, 12-lead electrocardiograms, physical examinations and virologic assessments, including viral load, viral tropism and CD4+ cell count determinations will be performed at the Screening visit and at regularly scheduled visits throughout the study. A blood sample will also be obtained and stored to potentially determine the genotype of the CCR5 receptor.

The primary objectives are:

1. Assess the safety and tolerability of 3 doses of INCB009471 or placebo when administered orally, once daily, as monotherapy for 14 days;
2. Determine the pharmacokinetics of 3 doses of INCB009471 or placebo when administered orally, once daily, as monotherapy for 14 days;
3. Evaluate the anti-retroviral activity of 3 doses of INCB009471 or placebo when administered orally, once daily, as monotherapy for 14 days

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic HIV-1 infected individuals that are treatmen naïve (ie less than 2 weeks prior ARV exposure) or treatment experienced subjects who are not currently on HAART and have not received any ARVs for 3 months prior to Screening.

* Males between 18 years and 65 years of age, utilizing adequate contraceptive methods.
* Post menopausal or surgically sterile females between 18 years and 65 years of age. Women of childbearing potential, utilizing adequate contraceptive methods.
* CD4-lymphocyte count >350 cells/mm3
* HIV-1 RNA copies/ml > 10,000.
* HIV-1 is CCR5 tropic virus only.
* CCR5 antagonist treatment naive.
* BMI > 16 to < 32 kg/m2.
* Have no clinically significant findings on screening evaluations, which in the opinion of the Investigator would interfere with the subject's ability to comply with the protocol.
* Able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

* Current or recent (<30 days) opportunistic infection.
* Presence of CXCR4- or dual-tropic HIV-1 virus at Screening or Baseline assessments.
* Subjects with chronic renal insufficiency
* Personal history of cardiac diseases.
* History or presence of an abnormal ECG.
* History of unstable ischemic heart disease or uncontrolled hypertension.
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* Subjects who have received radiation therapy or cytotoxic chemotherapeutic agents and have not recovered from side effects.
* Current treatment or treatment within 30 days or 5 half-lives with another investigational medication or current enrollment in another investigational drug protocol.
* Subjects with unstable medical condition (s), which , in the opinion of the Investigator would compromise their participation in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by monitoring adverse experiences. | Baseline, every 1-7 days following the initiation of treatment through Day 28 and then at Day 42 or the early study termination visit.

SECONDARY OUTCOMES:
The virological response to INCB009471 as monotherapy will be assessed by measuring HIV-1 RNA levels by the Roche Amplicor HIV-1 Monitor® Test, v1.5 - Quantitative. | Baseline, Days 4, 7, 10, 14, 16, 20 and 28 or the early termination study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Study Director — Incyte Corporation
Locations (6):
- United States (6):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Vero Beach, Florida
  - Boston, Massachusetts
  - Annandale, Virginia